CLINICAL TRIAL: NCT01521416
Title: The Cost of Illness Associated With Influenza in the UK
Brief Title: Cost of Illness Associated With Influenza in the UK
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 116313
Record Dates: First submitted 2012-01-26; First posted 2012-01-30 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: Influenza
Keywords: Illness; Influenza; Cost; UK
MeSH Terms: conditions — Influenza, Human | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cohort Group
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data of patients diagnosed with acute respiratory illness is extracted from General Practice Research Database (GPRD), Hospital Episode Statistics (HES), the Health Protection Agency (HPA), Office of National Statistics (ONS), and National Health Service (NHS) Reference Costs, during the period January 21st 2001 and March 31st 2009 inclusive.
  All analyses of primary care data (GPRD) and separately for secondary care (HES) data will be repeated for all eligible patients, and the subset of patients with a linkage to additional data (HES, ONS). All analysis including secondary care data will be restricted to the subset of patients with linked HES data. Estimates of average burden per patient and total burden in the UK will be performed. Burden is defined as both resource use and cost. Annual incidence and burden will be calculated.

SUMMARY:
The objective of this study is to describe the burden associated with influenza in the UK, from both primary and secondary care perspectives, and to stratify the burden by the annual degree of mismatch between predicted and actual virus strains.

DETAILED DESCRIPTION:
This is a retrospective, cross sectional, exploratory, observational study using database analysis and therefore there is no patient or user group involvement.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients coded within the database as having acute respiratory events that could be related to an infection between 2001 and 2009.
* Patients must have a minimum of 14 days observation before and after the index event to permit the capturing of complications attributable to influenza.

Exclusion Criteria:

Not Applicable

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients coded within the relevant database (GPRD and HES) as having acute respiratory events that could be related to an infection between 2001 and 2009.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Incidence of influenza-related events | Over the study time period (from January 21st 2001 to March 31st 2009 inclusive)
Number of confirmed influenza infections | Over the study time period (from January 21st 2001 to March 31st 2009 inclusive)
Assessment of resource use | Over the study time period (from January 21st 2001 to March 31st 2009 inclusive)
Evaluation of patient outcomes, treatments and costs (type and duration) | Over the study time period (from January 21st 2001 to March 31st 2009 inclusive)
Cause of deaths | Over the study time period (from January 21st 2001 to March 31st 2009 inclusive)
Incidence of influenza-related events in High Risk groups | Over the study time period (from January 21st 2001 to March 31st 2009 inclusive)
Incidence of complications and exacerbations | Over the study time period (from January 21st 2001 to March 31st 2009 inclusive)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline